CLINICAL TRIAL: NCT00973349
Title: A Pivotal Randomized, Single-Blind, Dose-Finding Study to Evaluate Immunogenicity, Safety and Tolerability of Different Formulations of an Adjuvanted and Non-Adjuvanted Egg-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Adult Subjects 18 or More Years of Age
Brief Title: Safety and Immunogenicity of A/H1N1-SOIV (Swine Flu) Vaccine With and Without Adjuvant in Non-Elderly and Elderly Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V112_01
Record Dates: First submitted 2009-09-02; First posted 2009-09-09 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Swine Flu; Flu; Vaccine; Adults; Elderly; Non-Elderly; Adjuvant
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- 3.75_(50)MF59 (Experimental): 50% of MF59 with 3.75 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 7.5 w/o MF59 (Experimental): 0% of MF59 with 7.5 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 7.5_(50)MF59 (Experimental): 50% of MF59 with 7.5 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 7.5_(100)MF59 (Experimental): 100% of MF59 with 7.5 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 15 w/o MF59 (Experimental): 0% of MF59 with 15 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 15_(50)MF59 (Experimental): 50% of MF59 with 15 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 15_(100)MF59 (Experimental): 100% of MF59 with 15 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f
- 30 w/o MF59 (Experimental): 0% of MF59 with 30 µg A/H1N1 antigen
  Interventions: Biological: MF59-eH1N1_f

INTERVENTIONS:
Biological: MF59-eH1N1_f — 8 arms consisting of different antigen combinations of A/H1N1 S-OIV and different percentages of MF59 adjuvant

SUMMARY:
This study will evaluate the safety and immunogenicity of different combinations of A/H1N1 S-OIV (swine flu) vaccine in non-elderly and elderly adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older in good health as determined by medical history, physical assessment and clinical judgement of the investigator and without influenza within the past 6 months.

Exclusion Criteria:

* History of serious disease.
* History of serious reaction following administration of vaccine or hypersensitivity to vaccine components.
* Known or suspected impairment/alteration of immune function.
* Receipt or planned receipt of seasonal trivalent influenza vaccine within 1 week before or after each study vaccination.
* Sexually active women of childbearing potential must use acceptable birth control during the treatment phase of the study.
* For additional entry criteria, please refer to protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2719 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccine and Diagnostics, Study Director — Novartis
Locations (21):
- United States (20):
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Meridien Clinical Research, Omaha, Nebraska
  - Regional Clinical Research, Endwell, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Triangle Medical Research Associates, Cary, North Carolina
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - Carolina Medical Trials, Winston-Salem, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - West Ridge Family Practice (adult), Erie, Pennsylvania
  - Primary Physicians Research Inc. (adult), Jefferson Hills, Pennsylvania
  - Omega Clinical Research, Warwick, Rhode Island
  - Research Across America, Dallas, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - J.Lewis Research, Inc./Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc./Foothill Family Clinic South, Salt Lake City, Utah
  - PI-Coor Clinical Research, Burke, Virginia
  - PI Coor Clinical Research, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Instituto Nacional de Ciencias, Tlalpan, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 21 sites in the US.
Groups:
- 3.75_(50)MF59 (18-64 Years); 3.75_(50)MF59 (≥ 65 Years): 50% of MF59 (an adjuvant) with 3.75 µg A/H1N1 antigen administered on day 1 and day 22
- 7.5 w/o MF59 (18-64 Years); 7.5 w/o MF59 (≥ 65 Years): 1 dose of 7.5 µg A/H1N1 administered on study day 1 and day 22
- 7.5_(50)MF59 (18-64 Years); 7.5_(50)MF59 (≥ 65 Years): 50% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen administered on study day 1 and day 22
- 7.5_(100)MF59 (18-64 Years); 7.5_(100)MF59 (≥ 65 Years): 100% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen administered on study day 1 and day 22
- 15 w/o MF59 (18-64 Years); 15 w/o MF59 (≥ 65 Years): 1 dose of 15 µg A/H1N1 administered on study day 1 and day 22
- 15_(50)MF59 (18-64 Years); 15_(50)MF59 (≥ 65 Years): 50% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen administered on study day 1 and day 22
- 15_(100)MF59 (18-64 Years); 15_(100)MF59 (≥ 65 Years): 100% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen administered on study day 1 and day 22
- 30 w/o MF59(18-64 Years); 30 w/o MF59(≥ 65 Years): 1 dose of 30 µg A/H1N1 administered on study day 1 and day 22
Period: Overall Study
Arm/Group | 3.75_(50)MF59 (18-64 Years) | 7.5 w/o MF59 (18-64 Years) | 7.5_(50)MF59 (18-64 Years) | 7.5_(100)MF59 (18-64 Years) | 15 w/o MF59 (18-64 Years) | 15_(50)MF59 (18-64 Years) | 15_(100)MF59 (18-64 Years) | 30 w/o MF59(18-64 Years) | 3.75_(50)MF59 (≥ 65 Years) | 7.5 w/o MF59 (≥ 65 Years) | 7.5_(50)MF59 (≥ 65 Years) | 7.5_(100)MF59 (≥ 65 Years) | 15 w/o MF59 (≥ 65 Years) | 15_(50)MF59 (≥ 65 Years) | 15_(100)MF59 (≥ 65 Years) | 30 w/o MF59(≥ 65 Years)
Started | 170 | 168 | 171 | 168 | 170 | 169 | 174 | 169 | 171 | 169 | 174 | 169 | 169 | 171 | 170 | 167
Completed | 166 | 165 | 166 | 163 | 165 | 165 | 172 | 166 | 167 | 163 | 174 | 167 | 168 | 171 | 168 | 165
Not Completed | 4 | 3 | 5 | 5 | 5 | 4 | 2 | 3 | 4 | 6 | 0 | 2 | 1 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Inappropriate enrolment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to classify | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population for immunology assessments. Participants from one center excluded for GCP issues.
Groups:
- 3.75_(50)MF59 (18 to 64): 50% of MF59 (an adjuvant) with 3.75 µg A/H1N1 antigen in subjects 18 to 64 years of age
- 7.5 w/o MF59 (18 to 64): 1 dose of 7.5 µg A/H1N1 in subjects 18 to 64 years of age
- 7.5_(50)MF59 (18 to 64): 50% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen in subjects 18 to 64 years of age
- 7.5_(100)MF59 (18 to 64): 100% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen in subjects 18 to 64 years of age
- 15 w/o MF59 (18 to 64): 1 dose of 15 µg A/H1N1 in subjects 18 to 64 years of age
- 15_(50)MF59 (18 to 64): 50% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen in subjects 18 to 64 years of age
- 15_(100)MF59 (18 to 64): 100% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen
- 30 w/o MF59 (18 to 64): 1 dose of 30 µg A/H1N1 in subjects 18 to 64 years of age
- 3.75_(50)MF59 (≥ 65 ): 50% of MF59 (an adjuvant) with 3.75 µg A/H1N1 antigen in subjects ≥ 65 years of age
- 7.5 w/o MF59 (≥ 65): 1 dose of 7.5 µg A/H1N1 in subjects ≥ 65 years of age
- 7.5_(50)MF59 (≥ 65): 50% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen in subjects ≥ 65 years of age
- 7.5_(100)MF59 (≥ 65): 100% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen in subjects ≥ 65 years of age
- 15 w/o MF59 (≥ 65): 1 dose of 15 µg A/H1N1 in subjects ≥ 65 years of age
- 15_(50)MF59 (≥ 65): 50% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen in subjects ≥ 65 years of age
- 15_(100)MF59 (≥ 65): 100% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen in subjects ≥ 65 years of age
- 30 w/o MF59 (≥ 65): 1 dose of 30 µg A/H1N1 in subjects ≥ 65 years of age
- Total: Total of all reporting groups
Arm/Group | 3.75_(50)MF59 (18 to 64) | 7.5 w/o MF59 (18 to 64) | 7.5_(50)MF59 (18 to 64) | 7.5_(100)MF59 (18 to 64) | 15 w/o MF59 (18 to 64) | 15_(50)MF59 (18 to 64) | 15_(100)MF59 (18 to 64) | 30 w/o MF59 (18 to 64) | 3.75_(50)MF59 (≥ 65 ) | 7.5 w/o MF59 (≥ 65) | 7.5_(50)MF59 (≥ 65) | 7.5_(100)MF59 (≥ 65) | 15 w/o MF59 (≥ 65) | 15_(50)MF59 (≥ 65) | 15_(100)MF59 (≥ 65) | 30 w/o MF59 (≥ 65) | Total
Number analyzed (Participants) | 155 | 153 | 157 | 153 | 155 | 154 | 159 | 154 | 170 | 168 | 172 | 168 | 168 | 171 | 169 | 166 | 2592
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.8) | 39.8 (12.9) | 39.1 (13.5) | 40.6 (12.2) | 41.8 (12.9) | 39.7 (13.1) | 38.8 (11.9) | 40.8 (13.0) | 70.8 (5.1) | 71.8 (5.6) | 71.4 (5.6) | 70.7 (5.1) | 71.0 (5.0) | 70.4 (4.9) | 71.3 (5.2) | 70.8 (5.3) | 39.6 (12.8)
Sex/Gender, Customized [Number; unit: participants]
  Male(18 to 64 or ≥65 years) | 61 | 62 | 57 | 59 | 57 | 69 | 71 | 63 | 54 | 88 | 71 | 70 | 68 | 74 | 79 | 76 | 1079
  Female(18 to 64 or ≥65 yrs) | 94 | 91 | 100 | 94 | 98 | 85 | 88 | 91 | 116 | 80 | 101 | 98 | 100 | 97 | 90 | 90 | 1513

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Results After Each Vaccination by Vaccine Group, in Participants 18 to 64 Years of Age
Description: Seroconversion is defined by CBER (Center for Biologics Evaluation, Research and Review) as the percentage of participants with either a prevaccination HI titer <1:10 and a post vaccination HI titer > 40 or a pre-vaccination HI titer > 10 and a minimum four-fold rise in post-vaccination HI antibody titer. Seroprotection is defined as participants having HI antibody titer ≥1:40.
Time Frame: 21 days after each vaccination
Population: The analysis was based on the per protocol population.
Measure: Number; unit: Participants
Groups:
- 3.75_(50)MF59: 50% of MF59 (an adjuvant) with 3.75 µg A/H1N1 antigen administered on day 1 and day 22
- 7.5 w/o MF59: 1 dose of 7.5 µg A/H1N1 administered on study day 1 and day 22
- 7.5_(50)MF59: 50% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen administered on study day 1 and day 22
- 7.5_(100)MF59: 100% of MF59 (an adjuvant) with 7.5 µg A/H1N1 antigen administered on study day 1 and day 22
- 15 w/o MF59: 1 dose of 15 µg A/H1N1 administered on study day 1 and day 22
- 15_(50)MF59: 50% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen administered on study day 1 and day 22
- 15_(100)MF59: 100% of MF59 (an adjuvant) with 15 µg A/H1N1 antigen administered on study day 1 and day 22
- 30 w/o MF59: 1 dose of 30 µg A/H1N1 administered on study day 1 and day 22
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 146 | 142 | 142 | 141 | 141 | 138 | 149 | 144
Participants
  Seroprotection Day 22 | 129 | 126 | 135 | 134 | 133 | 135 | 147 | 141
  Seroconversion Day 22 | 113 | 100 | 123 | 126 | 127 | 124 | 135 | 130
  Seroprotection Day 43 | 138 | 133 | 136 | 137 | 135 | 137 | 145 | 142
  Seroconversion Day 43 | 118 | 104 | 123 | 129 | 126 | 125 | 139 | 132
  Seroprotection Day 202 (N=79,65,78,80,73,74,74,76) | 68 | 51 | 67 | 70 | 56 | 59 | 65 | 69
  Seroconversion Day 202 (N=79,65,78,80,73,74,74,76) | 50 | 32 | 48 | 53 | 49 | 49 | 51 | 55
  Seroprotection Day 387(N=105,95,88,84,91,91,106,84 | 76 | 78 | 66 | 67 | 66 | 74 | 89 | 69
  Seroconversion Day387(N=105,95,88,84,91,91,106,84) | 52 | 48 | 50 | 53 | 58 | 62 | 71 | 54

2. Secondary Outcome: Geometric Mean HI Titer by Vaccine Groups; in Participants 18 to 64 Years of Age and ≥65 Years of Age
Description: Geometric mean hemagglutinin inhibition (HI) titer = GMT
Time Frame: 21 days after each vaccination
Population: The analysis was on the per protocol set. For this analysis, total subjects enrolled were stratified and randomized in two age groups, according to the CBER criteria, 18 to 64 years and over 64 years of age.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 296 | 289 | 306 | 289 | 300 | 293 | 303 | 294
Geometric Mean Titer
  Day 22(18-64yrs;N=146,142,142,141,141,138,149,144) | 299 [234 to 382] | 238 [185 to 306] | 379 [295 to 486] | 551 [429 to 708] | 536 [417 to 689] | 538 [418 to 693] | 677 [530 to 864] | 637 [497 to 817]
  Day 43(18-64yrs;N=146,142,142,141,141,138,149,144) | 327 [262 to 409] | 239 [198 to 299] | 359 [286 to 449] | 538 [429 to 675] | 412 [328 to 517] | 494 [393 to 621] | 618 [496 to 771] | 497 [397 to 622]
  Day 22 (≥65 yrs;N=150,147,164,148,159,155,154,150) | 138 [107 to 178] | 133 [103 to 172] | 146 [114 to 185] | 184 [143 to 238] | 187 [146 to 238] | 203 [159 to 261] | 252 [197 to 324] | 237 [184 to 305]
  Day 43 (≥65 yrs;N=150,147,164,148,159,155,154,150) | 135 [107 to 171] | 118 [93 to 149] | 131 [104 to 164] | 167 [132 to 212] | 151 [120 to 190] | 164 [130 to 207] | 240 [190 to 302] | 211 [167 to 267]
Statistical Analysis 1: Comparison: 3.75_(50)MF59 vs 7.5 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 1.265, 95% CI 2-sided [0.998 to 1.603] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 2: Comparison: 3.75_(50)MF59 vs 7.5_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.999, 95% CI 2-sided [0.791 to 1.262] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 3: Comparison: 3.75_(50)MF59 vs 7.5_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.708, 95% CI 2-sided [0.558 to 0.897] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 4: Comparison: 3.75_(50)MF59 vs 15 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.861, 95% CI 2-sided [0.681 to 1.089] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 5: Comparison: 3.75_(50)MF59 vs 15_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.754, 95% CI 2-sided [0.596 to 0.956] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 6: Comparison: 3.75_(50)MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.548, 95% CI 2-sided [0.434 to 0.693] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 7: Comparison: 3.75_(50)MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.646, 95% CI 2-sided [0.510 to 0.817] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 8: Comparison: 7.5 w/o MF59 vs 7.5_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at 43 = 0.790, 95% CI 2-sided [0.625 to 1.000] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 9: Comparison: 7.5 w/o MF59 vs 7.5_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at 43 = 0.560, 95% CI 2-sided [0.441 to 0.710] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 10: Comparison: 7.5 w/o MF59 vs 15 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at 43 = 0.681, 95% CI 2-sided [0.538 to 0.862] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 11: Comparison: 7.5 w/o MF59 vs 15_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at 43 = 0.597, 95% CI 2-sided [0.470 to 0.757] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 12: Comparison: 7.5 w/o MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.434, 95% CI 2-sided [0.342 to 0.549] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 13: Comparison: 7.5 w/o MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.511, 95% CI 2-sided [0.403 to 0.647] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 14: Comparison: 7.5_(50)MF59 vs 7.5_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.708, 95% CI 2-sided [0.560 to 0.896] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 15: Comparison: 7.5_(50)MF59 vs 15 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.862, 95% CI 2-sided [0.683 to 1.088] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 16: Comparison: 7.5_(50)MF59 vs 15_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.755, 95% CI 2-sided [0.597 to 0.954] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 17: Comparison: 7.5_(50)MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.549, 95% CI 2-sided [0.435 to 0.692] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 18: Comparison: 7.5_(50)MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.646, 95% CI 2-sided [0.511 to 0.817] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 19: Comparison: 7.5_(100)MF59 vs 15 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 1.217, 95% CI 2-sided [0.961 to 1.541] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 20: Comparison: 7.5_(100)MF59 vs 15_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 1.066, 95% CI 2-sided [0.841 to 1.352] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 21: Comparison: 7.5_(100)MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.775, 95% CI 2-sided [0.612 to 0.981] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 22: Comparison: 7.5_(100)MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.912, 95% CI 2-sided [0.719 to 1.157] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 23: Comparison: 15 w/o MF59 vs 15_(50)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.876, 95% CI 2-sided [0.692 to 1.109] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 24: Comparison: 15 w/o MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.637, 95% CI 2-sided [0.504 to 0.804] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 25: Comparison: 15 w/o MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.750, 95% CI 2-sided [0.593 to 0.949] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 26: Comparison: 15_(50)MF59 vs 15_(100)MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.727, 95% CI 2-sided [0.574 to 0.919] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 27: Comparison: 15_(50)MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 0.856, 95% CI 2-sided [0.675 to 1.084] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups
Statistical Analysis 28: Comparison: 15_(100)MF59 vs 30 w/o MF59; Two-sided 95% CI around the point estimates were to be presented for each endpoint; Test type: Non-Inferiority or Equivalence — The 2-sided CIs were examined against a non-inferiority margin of 0.67; Geometric mean ratio at day 43 = 1.178, 95% CI 2-sided [0.931 to 1.489] — Pairwise Comparisons of GMTs (95% CI) Between Vaccination Groups at Day 43, on the pooled age groups

3. Secondary Outcome: Number of Subjects With Seroconversion and With HI ≥1:40, in Participants 18 to 60 Years of Age
Description: Immunogenicity evaluation after each vaccination by vaccine group according to CHMP (Committee for Medicinal Products for Human Use) criteria. Seroconversion is defined as the percentage of participants with either a prevaccination HI titer <1:10 and a post vaccination HI titer > 40 or a pre-vaccination HI titer > 10 and a minimum four-fold rise in post-vaccination HI antibody titer. Seroprotection is defined as Hemagglutinin Inhibition (HI) antibody titer ≥1:40.
Time Frame: 21 days after each vaccination
Population: The analysis was on the per protocol set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 135 | 130 | 132 | 132 | 122 | 124 | 141 | 127
Participants
  Seroprotection Day 22 | 121 | 118 | 126 | 125 | 116 | 121 | 140 | 125
  Seroconversion Day 22 | 108 | 95 | 116 | 118 | 111 | 113 | 129 | 116
  Seroprotection Day 43 | 128 | 124 | 126 | 128 | 118 | 123 | 138 | 126
  Seroconversion Day 43 | 112 | 98 | 115 | 122 | 110 | 114 | 132 | 119

4. Primary Outcome: Immunogenicity Results After Each Vaccination by Vaccine Group, in Participants ≥65 Years of Age
Description: Seroconversion is defined by CBER as the percentage of participants with either a prevaccination HI titer <1:10 and a post vaccination HI titer > 40 or a pre-vaccination HI titer > 10 and a minimum four-fold rise in post-vaccination HI antibody titer. Seroprotection is defined as participants having HI antibody titer ≥1:40.
Time Frame: 21 days after each vaccination
Population: The analysis was on the per protocol set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 150 | 147 | 164 | 148 | 159 | 155 | 154 | 150
Participants
  Seroprotection Day 22 | 122 | 119 | 126 | 122 | 136 | 141 | 142 | 135
  Seroconversion Day 22 | 89 | 76 | 102 | 92 | 104 | 110 | 111 | 108
  Seroprotection Day 43 | 131 | 116 | 132 | 131 | 126 | 136 | 143 | 136
  Seroconversion Day 43 | 90 | 75 | 103 | 95 | 94 | 106 | 113 | 103
  Seroprotection Day 202 (N=80,71,85,79,84,82,87,82) | 54 | 41 | 45 | 52 | 55 | 45 | 63 | 57
  Seroconversion Day 202 (N=80,71,85,79,84,82,87,82) | 31 | 16 | 30 | 31 | 35 | 27 | 38 | 36
  Seroprotection Day 387(N=84,87,98,86,106,93,89,99) | 50 | 56 | 55 | 57 | 67 | 55 | 65 | 69
  Seroconversion Day 387(N=84,87,98,86,106,93,89,99) | 30 | 25 | 26 | 33 | 37 | 30 | 47 | 32

5. Secondary Outcome: Number of Subjects With Seroconversion and With HI ≥1:40, in Participants ≥61 Years of Age
Description: Immunogenicity evaluation after each vaccination by vaccine group according to CHMP criteria. Seroconversion is defined as the percentage of participants with either a prevaccination HI titer <1:10 and a post vaccination HI titer > 40 or a pre-vaccination HI titer > 10 and a minimum four-fold rise in post-vaccination HI antibody titer. Seroprotection is defined as Hemagglutinin Inhibition (HI) antibody titer ≥1:40.
Time Frame: 21 days after each vaccination
Population: The analysis was on the per protocol set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 161 | 159 | 174 | 157 | 178 | 169 | 162 | 167
Participants
  Seroprotection Day 22 | 130 | 127 | 135 | 131 | 153 | 155 | 149 | 151
  Seroconversion Day 22 | 94 | 81 | 109 | 100 | 120 | 121 | 117 | 122
  Seroprotection Day 43 | 140 | 125 | 142 | 140 | 143 | 150 | 150 | 152
  Seroconversion Day 43 | 96 | 81 | 111 | 102 | 110 | 117 | 120 | 116

6. Secondary Outcome: Geometric Mean Ratio From Baseline, in Participants 18 to 60 Years of Age and ≥61 Years of Age
Description: Immunogenicity evaluation after each vaccination by vaccine group according to CHMP criteria. Geometric Mean Ratio (GMR) of the hemagglutinin inhibition (HI)titers.
Time Frame: 21 days after vaccination
Population: The analysis was on the per protocol set. For this analysis, total subjects enrolled were stratified and randomized in two age groups, according to the CHMP criteria, 18 to 60 years and over 60 years of age.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Ratio
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 296 | 289 | 306 | 289 | 300 | 293 | 303 | 294
Geometric Mean Ratio
  Day 22 (18-60y; N=135,130,132,132,122,124,141,127) | 19 [15 to 26] | 15 [11 to 20] | 23 [17 to 31] | 33 [25 to 44] | 40 [30 to 54] | 36 [27 to 49] | 44 [33 to 58] | 47 [35 to 63]
  Day 43 (18-60y; N=135,130,132,132,122,124,141,127) | 20 [16 to 27] | 15 [11 to 20] | 22 [17 to 28] | 33 [25 to 43] | 31 [23 to 40] | 33 [25 to 44] | 40 [31 to 51] | 37 [28 to 48]
  Day 22 (≥61yrs; N=161,159,174,157,178,169,162,167) | 6.11 [4.8 to 7.78] | 4.65 [3.65 to 5.94] | 7.46 [5.91 to 9.41] | 8.63 [6.75 to 11] | 8.37 [6.64 to 11] | 9.6 [7.57 to 12] | 11 [9.04 to 15] | 10 [7.97 to 13]
  Day 43 (≥61 yrs;N=161,159,174,157,178,169,162,167) | 6.2 [4.97 to 7.75] | 4.18 [3.34 to 5.23] | 6.77 [5.47 to 8.4] | 7.78 [6.21 to 9.75] | 6.72 [5.43 to 8.31] | 7.78 [6.25 to 9.68] | 11 [8.76 to 14] | 8.8 [7.07 to 11]

7. Secondary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After the First Vaccination, in Participants 18 to 64 Years of Age
Description: Solicited local and systemic reactions that occurred within 7 days after the day of vaccination were used as indicators of reactogenicity.
Time Frame: 7 days after vaccination
Population: The population used in analysis was the safety set
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 169 | 168 | 170 | 165 | 170 | 168 | 173 | 168
Participants
  Pain | 67 | 38 | 51 | 78 | 27 | 57 | 78 | 44
  Erythema | 2 | 2 | 2 | 4 | 3 | 2 | 4 | 0
  Swelling | 9 | 6 | 4 | 6 | 4 | 3 | 13 | 3
  Induration | 11 | 5 | 9 | 9 | 8 | 8 | 15 | 7
  Tenderness | 63 | 44 | 59 | 79 | 42 | 64 | 89 | 51
  Chills | 6 | 9 | 11 | 8 | 9 | 8 | 14 | 10
  Myalgia | 29 | 22 | 28 | 29 | 21 | 30 | 37 | 24
  Arthralgia | 14 | 13 | 17 | 10 | 11 | 10 | 6 | 7
  Headache | 37 | 39 | 42 | 32 | 43 | 39 | 36 | 36
  Nausea | 14 | 15 | 19 | 8 | 12 | 13 | 16 | 13
  Vomiting (N=169, 168, 169, 165, 170, 168, 173,168) | 3 | 3 | 2 | 1 | 3 | 2 | 1 | 2
  Diarrhoea | 11 | 7 | 19 | 5 | 11 | 15 | 6 | 7
  Fatigue | 25 | 28 | 27 | 17 | 27 | 27 | 26 | 27
  Oral Temp. (≥40°C) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stay Home | 6 | 6 | 4 | 3 | 8 | 9 | 9 | 6

8. Secondary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After the Second Vaccination, in Participants 18 to 64 Years of Age
Description: as for outcome 7
Time Frame: 7 days after vaccination
Population: The analysis was on the safety set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 164 | 163 | 162 | 160 | 162 | 160 | 169 | 163
Participants
  Pain | 46 | 32 | 39 | 42 | 35 | 43 | 54 | 45
  Erythema (N=164,163,162,160,162,160,169,163) | 2 | 1 | 3 | 1 | 3 | 1 | 4 | 1
  Swelling (N=164,163,162,160,162,160,169,162) | 10 | 2 | 5 | 8 | 6 | 4 | 9 | 2
  Induration (N=164,163,162,160,162,160,169,163) | 7 | 5 | 6 | 7 | 5 | 11 | 13 | 11
  Tenderness (N=164,163,162,160,162,160,169,163) | 51 | 33 | 52 | 56 | 44 | 58 | 66 | 56
  Chills (N=164,163,162,160,162,160,169,163) | 9 | 3 | 4 | 5 | 5 | 7 | 5 | 2
  Myalgia (N=164,163,162,160,162,160,169,163) | 22 | 18 | 14 | 20 | 20 | 16 | 24 | 10
  Arthralgia (N=164,163,162,160,162,160,169,163) | 7 | 4 | 7 | 7 | 6 | 7 | 14 | 3
  Headache(N=164,163,162,160,162,160,169,163) | 28 | 17 | 26 | 23 | 25 | 32 | 26 | 17
  Nausea(N=164,163,162,160,162,160,169,163) | 5 | 7 | 9 | 8 | 4 | 9 | 13 | 6
  Vomiting (N=164,163,162,160,162,160,169,163) | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
  Diarrhoea(N=164,163,162,160,162,160,169,163) | 5 | 11 | 8 | 5 | 6 | 8 | 7 | 5
  Fatigue(N=164,163,162,160,162,160,169,163) | 17 | 12 | 15 | 18 | 12 | 18 | 26 | 10
  Oral Temp ≥40°C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stay Home (N=164,163,161,160,162,159,169,163) | 4 | 3 | 5 | 0 | 2 | 3 | 6 | 0
  Analg/antipyr (N=164,163,162,160,162,160,169,163) | 11 | 6 | 7 | 5 | 9 | 14 | 10 | 9

9. Secondary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After the First Vaccination, in Participants ≥65 Years of Age
Description: as for outcome 7
Time Frame: 7 days after vaccination
Population: The analysis was on the safety set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 170 | 166 | 173 | 169 | 169 | 171 | 169 | 167
Participants
  Pain | 18 | 8 | 22 | 30 | 15 | 27 | 16 | 19
  Erythema | 1 | 1 | 1 | 2 | 3 | 2 | 3 | 5
  Swelling | 1 | 6 | 2 | 14 | 1 | 1 | 1 | 10
  Induration | 8 | 8 | 5 | 10 | 2 | 6 | 7 | 14
  Tenderness | 27 | 10 | 23 | 42 | 24 | 28 | 39 | 32
  Chills | 6 | 8 | 5 | 4 | 6 | 1 | 5 | 3
  Myalgia | 20 | 14 | 19 | 21 | 17 | 15 | 21 | 14
  Arthralgia | 13 | 9 | 13 | 12 | 11 | 10 | 11 | 10
  Headache | 23 | 21 | 22 | 25 | 16 | 22 | 17 | 14
  Nausea | 2 | 4 | 2 | 3 | 6 | 5 | 6 | 7
  Vomitting (N=170,166,173,169.169,170,169,167) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Diarrhoea | 5 | 10 | 14 | 9 | 9 | 12 | 9 | 6
  Fatigue | 23 | 20 | 21 | 19 | 20 | 15 | 22 | 13
  Oral Temp ≥40°C | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Stay Home | 8 | 3 | 8 | 3 | 2 | 4 | 5 | 4
  Analg/antipyr (N=170,166,172,169.167,171,169,166) | 9 | 7 | 7 | 11 | 7 | 6 | 5 | 2

10. Secondary Outcome: Number of Participants Reporting Solicited Local and Systemic Reactions After the Second Vaccination, in Participants ≥65 Years of Age
Description: as for outcome 7
Time Frame: 7 days after vaccination
Population: The analysis was on the safety set.
Measure: Number; unit: Participants
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59
Number analyzed (Participants) | 164 | 156 | 171 | 160 | 166 | 168 | 165 | 165
Participants
  Pain (N=164,156,171,160,166,168,165,165) | 12 | 8 | 17 | 16 | 17 | 15 | 17 | 14
  Erythema (N=163,156,171,160,166,168,165,164) | 1 | 0 | 1 | 5 | 3 | 1 | 5 | 2
  Swelling (N=163,156,171,160,166,168,165,164) | 1 | 1 | 3 | 4 | 1 | 3 | 6 | 3
  Induration (N=163,156,171,160,166,168,165,164) | 3 | 3 | 7 | 4 | 2 | 6 | 7 | 6
  Tenderness (N=164,156,171,160,166,168,165,164) | 22 | 12 | 26 | 30 | 25 | 26 | 31 | 18
  Chills (N=163,156,171,160,166,168,165,164) | 2 | 7 | 7 | 4 | 5 | 3 | 5 | 3
  Myalgia (N=163,156,171,160,166,168,165,164) | 20 | 14 | 15 | 9 | 16 | 12 | 11 | 7
  Arthralgia (N=163,156,171,160,166,168,165,164) | 15 | 8 | 11 | 5 | 9 | 7 | 7 | 3
  Headache (N=163,156,171,160,166,168,165,164) | 14 | 13 | 17 | 12 | 15 | 10 | 11 | 10
  Nausea (N=163,156,171,160,166,168,165,164) | 4 | 5 | 5 | 3 | 7 | 4 | 4 | 2
  Vomiting (N=164,156,171,160,166,168,165,165) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
  Diarrhoea (N=163,156,171,160,166,168,165,164) | 4 | 5 | 10 | 2 | 6 | 6 | 6 | 2
  Fatigue (N=163,156,171,160,166,168,165,164) | 19 | 9 | 14 | 7 | 14 | 8 | 11 | 5
  Oral Temp≥40°C (N=164,156,171,160,166,168,165,165) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Stay Home(N=163,156,171,159,166,168,165,164) | 3 | 5 | 5 | 1 | 2 | 0 | 0 | 2
  Analg/antipyr (N=164,156,171,160,166,167,165,163) | 2 | 7 | 10 | 4 | 1 | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: All solicited AEs were collected for the first 3 weeks after each vaccination. SAEs, new onset of chronic diseases, AEs that led to withdrawal from study and AEs associated with medically attended visits, were collected for the whole study (days 1-387).
Description: A systematic AE is equivalent to an event that was solicited by the diary card, while a non-systematic event is equivalent to an event not solicited by the diary card. Safety was analyzed with data from all study centers; 10 enrolled participants were excluded for not receiving study vaccine or not providing safety data after first vaccination.
Groups:
- 3.75_(50)MF59; 3.75_(50)MF59 (Above 65 Yrs): 50% of MF59 with the lowest amount of A/H1N1 antigen
- 7.5 w/o MF59; 7.5 w/o MF59 (≥65 Yrs): 1 dose of 7.5 µg A/H1N1
- 15 w/o MF59; 15 w/o MF59 (≥ 65 Yrs): 1 dose of 15 µg A/H1N1
- 30 w/o MF59; 30 w/o MF59 (≥65 Yrs): 1 dose of 30 µg A/H1N1
- 7.5_(50)MF59 (≥65 Yrs): 50% of MF59 with 7.5 µg A/H1N1 antigen
- 7.5_(100)MF59 (≥65 Yrs): 100% of MF59 with 7.5 µg A/H1N1 antigen
- 15_(50)MF59 (≥65 Yrs): 50% of MF59 with 15 µg A/H1N1 antigen
- 15_(100)MF59 (≥65 Yrs): 100% of MF59 with 15 µg A/H1N1 antigen
Arm/Group | 3.75_(50)MF59 | 7.5 w/o MF59 | 7.5_(50)MF59 | 7.5_(100)MF59 | 15 w/o MF59 | 15_(50)MF59 | 15_(100)MF59 | 30 w/o MF59 | 3.75_(50)MF59 (Above 65 Yrs) | 7.5 w/o MF59 (≥65 Yrs) | 7.5_(50)MF59 (≥65 Yrs) | 7.5_(100)MF59 (≥65 Yrs) | 15 w/o MF59 (≥ 65 Yrs) | 15_(50)MF59 (≥65 Yrs) | 15_(100)MF59 (≥65 Yrs) | 30 w/o MF59 (≥65 Yrs)
Serious Adverse Events (participants affected / at risk) | 5/170 | 5/168 | 5/171 | 5/165 | 6/170 | 6/169 | 5/174 | 7/168 | 9/170 | 16/166 | 18/173 | 11/169 | 12/169 | 20/171 | 14/169 | 10/167
Other Adverse Events (participants affected / at risk) | 125/170 | 108/168 | 121/171 | 128/165 | 113/170 | 122/169 | 130/174 | 110/168 | 102/170 | 88/166 | 101/173 | 118/169 | 104/169 | 109/171 | 97/169 | 99/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3.75_(50)MF59 (N=170) | 7.5 w/o MF59 (N=168) | 7.5_(50)MF59 (N=171) | 7.5_(100)MF59 (N=165) | 15 w/o MF59 (N=170) | 15_(50)MF59 (N=169) | 15_(100)MF59 (N=174) | 30 w/o MF59 (N=168) | 3.75_(50)MF59 (Above 65 Yrs) (N=170) | 7.5 w/o MF59 (≥65 Yrs) (N=166) | 7.5_(50)MF59 (≥65 Yrs) (N=173) | 7.5_(100)MF59 (≥65 Yrs) (N=169) | 15 w/o MF59 (≥ 65 Yrs) (N=169) | 15_(50)MF59 (≥65 Yrs) (N=171) | 15_(100)MF59 (≥65 Yrs) (N=169) | 30 w/o MF59 (≥65 Yrs) (N=167)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Suicide Attempt (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder non-functioning (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis Reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penis Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneus Complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Resection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic Valve imcompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal Obstructuction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gallbladder Disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 3 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid Artery Occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ankle Operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive Emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
H1N1 Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3.75_(50)MF59 (N=170) | 7.5 w/o MF59 (N=168) | 7.5_(50)MF59 (N=171) | 7.5_(100)MF59 (N=165) | 15 w/o MF59 (N=170) | 15_(50)MF59 (N=169) | 15_(100)MF59 (N=174) | 30 w/o MF59 (N=168) | 3.75_(50)MF59 (Above 65 Yrs) (N=170) | 7.5 w/o MF59 (≥65 Yrs) (N=166) | 7.5_(50)MF59 (≥65 Yrs) (N=173) | 7.5_(100)MF59 (≥65 Yrs) (N=169) | 15 w/o MF59 (≥ 65 Yrs) (N=169) | 15_(50)MF59 (≥65 Yrs) (N=171) | 15_(100)MF59 (≥65 Yrs) (N=169) | 30 w/o MF59 (≥65 Yrs) (N=167)
Headache (Nervous system disorders) | 56 | 49 | 51 | 42 | 60 | 55 | 50 | 43 | 33 | 29 | 33 | 30 | 28 | 29 | 25 | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 8 | 7 | 8 | 8 | 6 | 8 | 4 | 3 | 2 | 7 | 4 | 4 | 5 | 5
Injection site pain (General disorders) | 97 | 68 | 90 | 109 | 72 | 102 | 112 | 80 | 42 | 23 | 42 | 60 | 51 | 57 | 50 | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 34 | 32 | 43 | 32 | 39 | 47 | 30 | 35 | 24 | 27 | 27 | 26 | 23 | 27 | 19
Fatigue (General disorders) | 33 | 33 | 35 | 31 | 31 | 37 | 36 | 31 | 36 | 24 | 29 | 23 | 26 | 19 | 28 | 17
Nausea (Gastrointestinal disorders) | 20 | 18 | 25 | 15 | 16 | 18 | 27 | 17 | 6 | 10 | 9 | 7 | 12 | 8 | 11 | 9
Diarrhoea (Gastrointestinal disorders) | 17 | 18 | 24 | 13 | 21 | 18 | 12 | 15 | 11 | 17 | 22 | 16 | 13 | 17 | 16 | 9
Injection site erythema (General disorders) | 23 | 15 | 21 | 14 | 15 | 11 | 23 | 13 | 15 | 12 | 15 | 22 | 16 | 14 | 23 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 17 | 22 | 22 | 22 | 16 | 19 | 13 | 29 | 18 | 21 | 23 | 16 | 17 | 21 | 14
Injection site induration (General disorders) | 15 | 9 | 15 | 13 | 12 | 14 | 20 | 17 | 11 | 11 | 11 | 10 | 5 | 10 | 15 | 20
Injection site swelling (General disorders) | 16 | 9 | 10 | 9 | 10 | 8 | 15 | 5 | 2 | 6 | 5 | 13 | 3 | 3 | 6 | 12
Chills (General disorders) | 15 | 13 | 15 | 12 | 13 | 15 | 15 | 11 | 8 | 12 | 10 | 8 | 9 | 4 | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 7 | 5 | 7 | 7 | 6 | 10 | 6 | 3 | 8 | 7 | 6 | 7 | 11 | 9
Nasopharyngitis (Infections and infestations) | 9 | 8 | 8 | 6 | 5 | 3 | 2 | 1 | 7 | 6 | 8 | 10 | 4 | 6 | 7 | 5
Sinusitis (Infections and infestations) | 8 | 6 | 19 | 11 | 16 | 7 | 6 | 13 | 8 | 9 | 13 | 9 | 9 | 8 | 5 | 7
Upper Respiratory Tract infection (Infections and infestations) | 4 | 14 | 9 | 11 | 8 | 9 | 13 | 6 | 7 | 9 | 5 | 14 | 7 | 6 | 8 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 3 | 3 | 1 | 1 | 0 | 12 | 4 | 0 | 5 | 6 | 3 | 1 | 6
Bronchitis (Infections and infestations) | 3 | 10 | 4 | 6 | 7 | 5 | 3 | 5 | 4 | 4 | 6 | 3 | 5 | 5 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No